CLINICAL TRIAL: NCT01362010
Title: Pilot, Multicenter, Randomized, Double Blind, Placebo Controlled, Parallel Group, Dose Range Finding Study, to Evaluate the Tolerability and Safety of FXFM244 Antibiotic Foam and to Monitor Its Clinical Effect in Acne Vulgaris Patients
Brief Title: Clinical Study to Evaluate Tolerability and Safety of FXFM244 and to Monitor Clinical Effect in Acne Vulgaris Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vyne Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FX2010-03
Record Dates: First submitted 2011-05-26; First posted 2011-05-27 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2013-08

CONDITIONS: Acne Vulgaris
Keywords: Acne; Acne Vulgaris; Topical; Minocycline; Foam; Phase II
MeSH Terms: conditions — Acne Vulgaris; cyclopia sequence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Topical Minocycline Foam FXFM244 - 4% (Experimental): Active ingredient: Minocycline Concentration: 4% Route: Topical Dosage schedule: Once daily, evening.
  Interventions: Drug: Topical Minocycline Foam FXFM244
- Topical Minocycline Foam FXFM244 - 1% (Experimental): Active ingredient: Minocycline Concentration: 1% Route: Topical Dosage schedule: Once daily, evening.
  Interventions: Drug: Topical Minocycline Foam FXFM244
- Placebo foam (Placebo Comparator): Active ingredient: None Route: Topical Dosage schedule: Once daily, evening
  Interventions: Drug: Topical Minocycline Foam FXFM244

INTERVENTIONS:
Drug: Topical Minocycline Foam FXFM244 — Topically applied once a day.
  Other Names: FXFM244 antibiotic foam

SUMMARY:
The purpose of this study is to evaluate the tolerability and safety and to determine whether FXFM244 Antibiotic Foam is effective in the treatment of Acne Vulgaris.

DETAILED DESCRIPTION:
This is a phase IIa prospective, multicenter, randomized, double blind, placebo controlled, parallel group, dose range finding clinical study to evaluate the safety, tolerability and efficacy of Minocycline Foam 1% and 4% for the treatment of Acne Vulgaris.

The study consists of a screening / baseline visit, a treatment period where patients will be treated topically on the facial skin areas affected by acne twice daily for 12 weeks, followed by a post-treatment follow up visit 4 weeks after end of treatment. The first dose will be applied in the presence of the study investigator or his assignee. Subsequent applications will be made by the patients.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of Acne Vulgaris with facial involvement.
* A minimum of 20 but not more than 50 inflammatory lesions on the face (papules and/ or pustules).
* A minimum of 25 but not more than 100 non-inflammatory lesions on the face (opened and/or closed comedones).
* No significant nodulocystic acne on the face (≤ 2 lesions).
* A score of >3 (Moderate) on the Investigator's Global Assessment Scale.
* Patient is male or female between the ages of 12 to 25.
* No known medical conditions that, in the Investigator's opinion could interfere with study participation.
* Patient is willing to refrain from use of all other topical acne medications or antibiotics during the study.
* Patient is willing to refrain from use of moisturizers, new brands of make-up, creams, lotions, powders or any topical product other than the assigned treatment to the treatment area.
* Patient is willing and able to comply with all requirement of the protocol.
* Patient is willing and able to give written informed consent prior to participation in the study.
* If female of childbearing potential, willing to use an acceptable form of birth control during the study. Use of oral contraceptives must remain constant within 3 month prior to baseline and throughout the study.

Exclusion Criteria:

* Acne Conglobata, Acne Fulminas, secondary acne (chloracne, drug induced acne), or severe acne requiring systemic treatment.
* Presence of any facial skin condition that would interfere with the diagnosis or assessment of Acne Vulgaris (e.g. rosacea, dermatitis, psoriasis, squamos cell carcinoma, eczema, acneform eruptions caused by medications, steroid acne, steroid folliculitis, or bacterial folliculitis).
* Excessive facial hair (beards, sideburns, moustaches, etc.) that would interfere with diagnosis or assessment of Acne Vulgaris.
* Known or suspected hypersensitivity to Minocycline or any of the excipients in the Study Medication.
* Concomitant medication:
* Use within 6 month prior to baseline of topical retinoids, oral retinoids (Accutane®) or therapeutic Protocol No. FX2010-03 Foamix Ltd. Page 8 of 28 Confidential Ver: 02 Oct-31-2011 vitamin A supplements of greater than 10,000 units/day (multivitamins are allowed).
* Use of systemic steroids, systemic antibiotics, systemic treatment for Acne Vulgaris, systemic antiinflammatory agents within 4 weeks prior to baseline.
* Use of topical steroids, α-hydroxy/glycolic acid, benzoyl peroxide, topical antibiotics, topical treatment for Acne Vulgaris, topical anti-inflammatory agents within 2 weeks prior to baseline.
* Use for less than 3 month prior to baseline of estrogens or change in oral contraceptives therapy within less than 3 month prior to baseline;
* Use on the face of: cryodestruction or chemodestruction, dermabrasion, photodynamic therapy, acne surgery, intralesional steroids or X-ray therapy within 4 weeks prior to baseline..
* Alcohol or drug abuse, according to assessment by the investigator.
* Use of another investigational drug within 30 days prior to baseline.
* Pregnant or lactating women.
* Use of tanning booths, sunbathing, or excessive exposure to the sun should be prohibited during the study.
* Participation in clinical trial in the previous month.

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Actual)
Dates: Start 2012-01; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Decrease in lesions count | 12 weeks
  The change in lesion count (inflammatory, non-inflammatory, and total) after 12 weeks of treatment compared to baseline
Investigator global assessment | 12 weeks
  Physician's Global Improvement Assessment

SECONDARY OUTCOMES:
% change in lesions count | 12 weeks
  The % change in lesions count (inflammatory, non-inflammatory, and total) after 12 weeks of treatment compared to baseline
Global assessment of improvement by photographs | 12 weeks
  The photographs will assist in comparison of efficacy at subsequent visits compared to baseline
Subject-reported outcome assessment | 12 weeks
Subjects safety | 12 weeks
  safety parameters will be assessed by
  * Physical examination
  * Vital signs (HR, BP, Body temperature)
  * Adverse events recording
  * Clinical assessment of skin irritation

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Shiri, Prof., Principal Investigator — Clalit Health Services; Eli Sprecher, MD, Principal Investigator — Sourasky Medical Center; Avner Shemer, Prof., Principal Investigator — Lev Yasmin clinic, Netanya, Israel
Locations (3):
- Israel (3):
  - Lev Yasmin clinic, Netanya
  - Sourasky medical center, Tel Aviv
  - Tel-Nordau Clalit health services, Tel Aviv